CLINICAL TRIAL: NCT00876447
Title: A Long-term Follow-up Study of Botulinum Toxin Type A in Patients With Overactive Bladder as a Result of Spinal Injury or Multiple Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 191622-094
Record Dates: First submitted 2009-04-01; First posted 2009-04-06 (Estimated); Results first posted 2014-06-13 (Estimated); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botulinum Toxin Type A 300U (Experimental): Botulinum toxin Type A 300U injections into the detrusor > 12 weeks as needed for up to 3 years.
  Interventions: Biological: Botulinum Toxin Type A 300U
- Botulinum Toxin Type A 200U (Experimental): Botulinum toxin Type A 200U injections into the detrusor > 12 weeks as needed for up to 3 years.
  Interventions: Biological: Botulinum Toxin Type A 200U

INTERVENTIONS:
Biological: Botulinum Toxin Type A 300U — Botulinum toxin Type A 300U injections into the detrusor > 12 weeks as needed for up to 3 years.
  Other Names: BOTOX®
  Arms: Botulinum Toxin Type A 300U
Biological: Botulinum Toxin Type A 200U — Botulinum toxin Type A 200U injections into the detrusor > 12 weeks as needed for up to 3 years.
  Other Names: BOTOX®
  Arms: Botulinum Toxin Type A 200U

SUMMARY:
The purpose of this study is to assess the long-term safety and effectiveness of botulinum toxin type A on patients with overactive bladder as a result of spinal cord injury or multiple sclerosis. This is a follow-up study to two Allergan sponsored studies (NCT00311376 and NCT00461292).

DETAILED DESCRIPTION:
Botulinum toxin Type A 300U has been discontinued from the study. Patients remaining in the arm containing botulinum toxin Type A 300U will receive botulinum toxin Type A 200U moving forward. Also, the masking of the study is now open-label.

ELIGIBILITY:
Inclusion Criteria:

* Patient has participated in study 191622-515 or 191622-516 and the following criteria fulfilled:

  * Patient completed at least 52 weeks in the preceding study.
  * No longer than 6 months has elapsed since completion of the preceding study
  * Patient has not received any prohibited medications during any intervening period between the preceding study and this long-term study.

Exclusion Criteria:

* History or evidence of pelvic or urologic abnormality.
* Previous or current diagnosis of bladder or prostate cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 397 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2013-06-12 (Actual); Study Completion 2013-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (22):
- Middlebury, Connecticut, United States
- Randwick, Australia
- Innsbruck, Austria
- Ghent, Belgium
- Rio de Janeiro, Brazil
- Victoria, British Columbia, Canada
- Ostrava, Czechia
- Salouël, France
- Kiel, Germany
- Florence, Italy
- Amsterdam, Netherlands
- Epsom, New Zealand
- Poznan, Poland
- Porto, Portugal
- Moscow, Russia
- Singapore, Singapore
- Prešov, Slovakia
- Pretoria, South Africa
- Santa Cruz de Tenerife, Spain
- Hualien City, Taiwan
- Kiev, Ukraine
- London, United Kingdom

REFERENCES:
- [Background] Kennelly M, Dmochowski R, Schulte-Baukloh H, Ethans K, Del Popolo G, Moore C, Jenkins B, Guard S, Zheng Y, Karsenty G; 191622-094 Investigators. Efficacy and safety of onabotulinumtoxinA therapy are sustained over 4 years of treatment in patients with neurogenic detrusor overactivity: Final results of a long-term extension study. Neurourol Urodyn. 2017 Feb;36(2):368-375. doi: 10.1002/nau.22934. Epub 2015 Nov 24. PMID 26607743

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a long-term follow-up study that enrolled patients after participation in Study 191622-515 or 191622-516. A total of 397 patients were enrolled and 388 patients received at least 1 BOTOX treatment in study 191622-094 or in the preceding studies.
Pre-assignment Details: The protocol was amended to remove the 300 U dose. Patients ongoing in the study who were treated with 300 U BOTOX prior to the amendment were assigned to 200 U BOTOX for all subsequent treatments. Participant Flow and Baseline Characteristics are based on the first BOTOX dose that patients received.
Period: Overall Study
Arm/Group | Botulinum Toxin Type A 300U | Botulinum Toxin Type A 200U
Started | 185 | 203
Completed | 105 | 122
Not Completed | 80 | 81
Not completed — Other miscellaneous reasons | 3 | 8
Not completed — Site closure | 19 | 14
Not completed — Protocol Violation | 9 | 3
Not completed — Personal reasons | 30 | 28
Not completed — Lost to Follow-up | 6 | 15
Not completed — Pregnancy | 4 | 2
Not completed — Lack of Efficacy | 5 | 3
Not completed — Adverse Event | 4 | 8

BASELINE CHARACTERISTICS:
Population: BOTOX-Treated population includes all patients who enrolled in this study and who received at least one BOTOX treatment, regardless of which study they received it in (study 191622-094 or their preceding study 191622-515 or 191622-516). The treatment groups are based on the first BOTOX dose that patients received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Botulinum Toxin Type A 300U | Botulinum Toxin Type A 200U | Total
Number analyzed (Participants) | 185 | 203 | 388
Age, Customized [Count of Participants; unit: Participants]
  <40 years | 55 | 57 | 112
  ≥40 to 64 years | 116 | 135 | 251
  ≥65 to 74 years | 14 | 10 | 24
  ≥75 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 118 | 234
  Male | 69 | 85 | 154

OUTCOME MEASURES:

1. Primary Outcome: Change From Study Baseline in the Daily Average Number of Urinary Incontinence Episodes
Description: Urinary incontinence is defined as involuntary loss of urine as recorded in a patient bladder diary in the 3 consecutive days prior to each study visit for study 191622-094 (or 7 days prior to each visit in study 191622-515 or 191622-516). The number of incontinence episodes are averaged daily during this period. The initial study baseline is obtained from the patient bladder diary in the 7 consecutive days prior to the first treatment in either study 191622-515 or 191622-516. A negative number change from baseline indicates a reduction in incontinence episodes (improvement).
Time Frame: Study Baseline, Week 6 Treatment Cycle 1
Population: BOTOX-Treated Population: all patients with data at the time point who received at least 1 BOTOX treatment since the start of their clinical study participation (in study 191622-094, 191622-515 or 191622-516); analyses are based on actual treatment received
Measure: Mean (Standard Deviation); unit: Incontinence Episodes
Arm/Group | Botulinum Toxin Type A 300U | Botulinum Toxin Type A 200U
Number analyzed (Participants) | 183 | 201
Incontinence Episodes
  Study Baseline (BL) | 4.4 (2.54) | 4.5 (2.64)
  Chg from Study BL at Wk 6 Tmt Cycle1 (N=176, 195) | -3.4 (3.16) | -3.2 (2.69)

2. Primary Outcome: Change From Study Baseline in the Daily Average Number of Urinary Incontinence Episodes
Description: as for outcome 1
Time Frame: Study Baseline, Week 6 Treatment Cycle 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Incontinence Episodes
Arm/Group | Botulinum Toxin Type A 300U | Botulinum Toxin Type A 200U
Number analyzed (Participants) | 161 | 186
Incontinence Episodes
  Study Baseline | 4.5 (2.62) | 4.6 (2.71)
  Chg from Study BL at Wk 6 Tmt Cycle2 (N=153, 175) | -3.5 (3.13) | -3.3 (2.85)

3. Primary Outcome: Change From Study Baseline in the Daily Average Number of Urinary Incontinence Episodes
Description: as for outcome 1
Time Frame: Study Baseline, Week 6 Treatment Cycle 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Incontinence Episodes
Arm/Group | Botulinum Toxin Type A 300U | Botulinum Toxin Type A 200U
Number analyzed (Participants) | 118 | 173
Incontinence Episodes
  Study Baseline | 4.4 (2.33) | 4.6 (2.65)
  Chg from Study BL at Wk 6 Tmt Cycle3 (N=109, 164) | -3.3 (2.39) | -3.5 (2.96)

4. Primary Outcome: Change From Study Baseline in the Daily Average Number of Urinary Incontinence Episodes
Description: as for outcome 1
Time Frame: Study Baseline, Week 6 Treatment Cycle 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Incontinence Episodes
Arm/Group | Botulinum Toxin Type A 300U | Botulinum Toxin Type A 200U
Number analyzed (Participants) | 67 | 149
Incontinence Episodes
  Study Baseline | 4.4 (2.13) | 4.4 (2.57)
  Chg from Study BL at Wk 6 Tmt Cycle4 (N=62, 141) | -3.4 (2.57) | -3.5 (2.61)

5. Primary Outcome: Change From Study Baseline in the Daily Average Number of Urinary Incontinence Episodes
Description: as for outcome 1
Time Frame: Study Baseline, Week 6 Treatment Cycle 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Incontinence Episodes
Arm/Group | Botulinum Toxin Type A 300U | Botulinum Toxin Type A 200U
Number analyzed (Participants) | 33 | 108
Incontinence Episodes
  Study Baseline | 4.1 (2.34) | 4.6 (2.57)
  Chg from Study BL at Wk 6 Tmt Cycle5 (N=29, 99) | -3.7 (2.82) | -3.6 (2.27)

6. Secondary Outcome: Change From Study Baseline in the Incontinence Quality of Life Instrument (I-QOL) Total Summary Score
Description: The I-QOL questionnaire is a validated, disease-specific quality of life (QOL) questionnaire containing 22 questions designed to measure the impact of urinary incontinence on patients' lives. Each question is answered on a 5-point scale (1 = worst QOL and 5 = best QOL). The scores are totaled over the 22 questions and normalized to a score of 0-100 (0 = worst QOL and 100= best QOL). The I-QOL total score is calculated by combining the 22-item subscores from the 3 I-QOL domains: Avoidance Limiting Behavior, Psychological Impact, and Social Embarrassment. The initial study baseline is obtained from data collected prior to the first treatment in Study 191622-515 or 191622-516. Positive number changes from baseline indicate improved QOL.
Time Frame: Study Baseline, Week 6 Treatment Cycle 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Botulinum Toxin Type A 300U | Botulinum Toxin Type A 200U
Number analyzed (Participants) | 185 | 202
Scores on a Scale
  Study Baseline | 33.9 (18.19) | 34.4 (18.18)
  Chg from Study BL at Wk 6 Tmt Cycle1 (N=180, 199) | 32.3 (26.07) | 30.3 (26.37)

7. Secondary Outcome: Change From Study Baseline in the Incontinence Quality of Life Instrument (I-QOL) Total Summary Score
Description: as for outcome 6
Time Frame: Study Baseline, Week 6 Treatment Cycle 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Botulinum Toxin Type A 300U | Botulinum Toxin Type A 200U
Number analyzed (Participants) | 162 | 185
Scores on a Scale
  Study Baseline | 33.3 (18.17) | 33.8 (18.17)
  Chg from Study BL at Wk 6 Tmt Cycle2 (N=157, 178) | 31.4 (27.73) | 33.5 (26.23)

8. Secondary Outcome: Change From Study Baseline in the Incontinence Quality of Life Instrument (I-QOL) Total Summary Score
Description: as for outcome 6
Time Frame: Study Baseline, Week 6 Treatment Cycle 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Botulinum Toxin Type A 300U | Botulinum Toxin Type A 200U
Number analyzed (Participants) | 118 | 173
Scores on a Scale
  Study Baseline | 32.5 (17.83) | 34.8 (18.95)
  Chg from Study BL at Wk 6 Tmt Cycle3 (N=114, 164) | 28.8 (28.96) | 30.4 (29.25)

9. Secondary Outcome: Change From Study Baseline in the Incontinence Quality of Life Instrument (I-QOL) Total Summary Score
Description: as for outcome 6
Time Frame: Study Baseline, Week 6 Treatment Cycle 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Botulinum Toxin Type A 300U | Botulinum Toxin Type A 200U
Number analyzed (Participants) | 66 | 151
Scores on a Scale
  Study Baseline | 27.9 (16.66) | 35.5 (17.70)
  Chg from Study BL at Wk 6 Tmt Cycle4 (N=63, 147) | 30.4 (31.77) | 30.1 (26.07)

10. Secondary Outcome: Change From Study Baseline in the Incontinence Quality of Life Instrument (I-QOL) Total Summary Score
Description: as for outcome 6
Time Frame: Study Baseline, Week 6 Treatment Cycle 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Botulinum Toxin Type A 300U | Botulinum Toxin Type A 200U
Number analyzed (Participants) | 31 | 109
Scores on a Scale
  Study Baseline | 32.0 (16.13) | 33.0 (19.61)
  Chg from Study BL at Wk 6 Tmt Cycle5 (N=28, 100) | 36.6 (28.28) | 27.1 (24.54)

11. Secondary Outcome: Change From Study Baseline in Volume Per Void
Description: The total volume voided (voluntary or by catheterization) is recorded by the patient over a 24-hour period preceding the study visit. The average volume per voiding episode is derived by dividing the total volume collected in a 24-hour period by the total number of urinary episodes with volume recorded in the same 24-hour period. The initial study baseline is obtained from data collected prior to the first treatment in Study 191622-515 or 191622-516. Positive number changes from baseline indicate improvement.
Time Frame: Study Baseline, Week 6 Treatment Cycle 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Milliliters (mL)
Arm/Group | Botulinum Toxin Type A 300U | Botulinum Toxin Type A 200U
Number analyzed (Participants) | 178 | 196
Milliliters (mL)
  Study Baseline | 147.3 (90.15) | 154.2 (96.54)
  Chg from Study BL at Wk 6 Tmt Cycle1 (N=168, 186) | 133.8 (137.23) | 133.2 (128.19)

12. Secondary Outcome: Change From Study Baseline in Volume Per Void
Description: as for outcome 11
Time Frame: Study Baseline, Week 6 Treatment Cycle 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Milliliters (mL)
Arm/Group | Botulinum Toxin Type A 300U | Botulinum Toxin Type A 200U
Number analyzed (Participants) | 157 | 181
Milliliters (mL)
  Study Baseline | 149.8 (91.03) | 151.9 (95.22)
  Chg from Study BL at Wk 6 Tmt Cycle2 (N=146, 168) | 148.0 (134.45) | 135.1 (127.62)

13. Secondary Outcome: Change From Study Baseline in Volume Per Void
Description: as for outcome 11
Time Frame: Study Baseline, Week 6 Treatment Cycle 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Milliliters (mL)
Arm/Group | Botulinum Toxin Type A 300U | Botulinum Toxin Type A 200U
Number analyzed (Participants) | 114 | 168
Milliliters (mL)
  Study Baseline | 155.0 (90.70) | 149.6 (91.12)
  Chg from Study BL at Wk 6 Tmt Cycle3 (N=105, 158) | 166.9 (133.59) | 157.5 (129.81)

14. Secondary Outcome: Change From Study Baseline in Volume Per Void
Description: as for outcome 11
Time Frame: Study Baseline, Week 6 Treatment Cycle 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Milliliters (mL)
Arm/Group | Botulinum Toxin Type A 300U | Botulinum Toxin Type A 200U
Number analyzed (Participants) | 65 | 143
Milliliters (mL)
  Study Baseline | 159.7 (89.37) | 151.7 (93.65)
  Chg from Study BL at Wk 6 Tmt Cycle4 (N=61, 135) | 170.8 (128.26) | 147.3 (122.09)

15. Secondary Outcome: Change From Study Baseline in Volume Per Void
Description: as for outcome 11
Time Frame: Study Baseline, Week 6 Treatment Cycle 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Milliliters (mL)
Arm/Group | Botulinum Toxin Type A 300U | Botulinum Toxin Type A 200U
Number analyzed (Participants) | 32 | 104
Milliliters (mL)
  Study Baseline | 182.7 (85.03) | 140.8 (91.32)
  Chg from Study BL at Wk 6 Tmt Cycle5 (N=28, 95) | 163.5 (106.44) | 160.2 (119.40)

ADVERSE EVENTS:
Description: The Botox-Treated Population includes all patients who received at least 1 BOTOX treatment (in Study 191622-094, 191622-515 or 191622-516) and is used to assess adverse events (AEs) and serious adverse events (SAEs). AEs and SAEs are reported by treatment cycle.
Groups:
- Botulinum Toxin Type A 300U Treatment Cycle 1; Botulinum Toxin Type A 300U Treatment Cycle 2; Botulinum Toxin Type A 300U Treatment Cycle 3; Botulinum Toxin Type A 300U Treatment Cycle 4; Botulinum Toxin Type A 300U Treatment Cycle 5; Botulinum Toxin Type A 300U Treatment Cycle 6; Botulinum Toxin Type A 300U Treatment Cycle 7; Botulinum Toxin Type A 300U Treatment Cycle 8; Botulinum Toxin Type A 300U Treatment Cycle 9; Botulinum Toxin Type A 300U Treatment Cycle 10; Botulinum Toxin Type A 300U Treatment Cycle 11; Botulinum Toxin Type A 300U Treatment Cycle 12; Botulinum Toxin Type A 300U Treatment Cycle 13: Botulinum toxin Type A 300U injections into the detrusor > 12 weeks for up to 3 years.
- Botulinum Toxin Type A 200U Treatment Cycle 1; Botulinum Toxin Type A 200U Treatment Cycle 2; Botulinum Toxin Type A 200U Treatment Cycle 3; Botulinum Toxin Type A 200U Treatment Cycle 4; Botulinum Toxin Type A 200U Treatment Cycle 5; Botulinum Toxin Type A 200U Treatment Cycle 6; Botulinum Toxin Type A 200U Treatment Cycle 7; Botulinum Toxin Type A 200U Treatment Cycle 8; Botulinum Toxin Type A 200U Treatment Cycle 9; Botulinum Toxin Type A 200U Treatment Cycle 10; Botulinum Toxin Type A 200U Treatment Cycle 11; Botulinum Toxin Type A 200U Treatment Cycle 12; Botulinum Toxin Type A 200U Treatment Cycle 13: Botulinum toxin Type A 200U injections into the detrusor > 12 weeks as needed for up to 3 years.
Arm/Group | Botulinum Toxin Type A 300U Treatment Cycle 1 | Botulinum Toxin Type A 200U Treatment Cycle 1 | Botulinum Toxin Type A 300U Treatment Cycle 2 | Botulinum Toxin Type A 200U Treatment Cycle 2 | Botulinum Toxin Type A 300U Treatment Cycle 3 | Botulinum Toxin Type A 200U Treatment Cycle 3 | Botulinum Toxin Type A 300U Treatment Cycle 4 | Botulinum Toxin Type A 200U Treatment Cycle 4 | Botulinum Toxin Type A 300U Treatment Cycle 5 | Botulinum Toxin Type A 200U Treatment Cycle 5 | Botulinum Toxin Type A 300U Treatment Cycle 6 | Botulinum Toxin Type A 200U Treatment Cycle 6 | Botulinum Toxin Type A 300U Treatment Cycle 7 | Botulinum Toxin Type A 200U Treatment Cycle 7 | Botulinum Toxin Type A 300U Treatment Cycle 8 | Botulinum Toxin Type A 200U Treatment Cycle 8 | Botulinum Toxin Type A 300U Treatment Cycle 9 | Botulinum Toxin Type A 200U Treatment Cycle 9 | Botulinum Toxin Type A 300U Treatment Cycle 10 | Botulinum Toxin Type A 200U Treatment Cycle 10 | Botulinum Toxin Type A 300U Treatment Cycle 11 | Botulinum Toxin Type A 200U Treatment Cycle 11 | Botulinum Toxin Type A 300U Treatment Cycle 12 | Botulinum Toxin Type A 200U Treatment Cycle 12 | Botulinum Toxin Type A 300U Treatment Cycle 13 | Botulinum Toxin Type A 200U Treatment Cycle 13
Serious Adverse Events (participants affected / at risk) | 28/185 | 35/203 | 26/163 | 21/187 | 20/119 | 19/175 | 11/69 | 20/153 | 5/34 | 11/110 | 0/16 | 9/70 | 0/8 | 6/48 | 0/0 | 0/36 | 0/0 | 2/22 | 0/0 | 1/11 | 0/0 | 0/5 | 0/0 | 0/2 | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 154/185 | 170/203 | 126/163 | 147/187 | 89/119 | 123/175 | 51/69 | 109/153 | 19/34 | 72/110 | 8/16 | 46/70 | 3/8 | 28/48 | 0/0 | 23/36 | 0/0 | 13/22 | 0/0 | 5/11 | 0/0 | 3/5 | 0/0 | 1/2 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Botulinum Toxin Type A 300U Treatment Cycle 1 (N=185) | Botulinum Toxin Type A 200U Treatment Cycle 1 (N=203) | Botulinum Toxin Type A 300U Treatment Cycle 2 (N=163) | Botulinum Toxin Type A 200U Treatment Cycle 2 (N=187) | Botulinum Toxin Type A 300U Treatment Cycle 3 (N=119) | Botulinum Toxin Type A 200U Treatment Cycle 3 (N=175) | Botulinum Toxin Type A 300U Treatment Cycle 4 (N=69) | Botulinum Toxin Type A 200U Treatment Cycle 4 (N=153) | Botulinum Toxin Type A 300U Treatment Cycle 5 (N=34) | Botulinum Toxin Type A 200U Treatment Cycle 5 (N=110) | Botulinum Toxin Type A 300U Treatment Cycle 6 (N=16) | Botulinum Toxin Type A 200U Treatment Cycle 6 (N=70) | Botulinum Toxin Type A 300U Treatment Cycle 7 (N=8) | Botulinum Toxin Type A 200U Treatment Cycle 7 (N=48) | Botulinum Toxin Type A 300U Treatment Cycle 8 (N=0) | Botulinum Toxin Type A 200U Treatment Cycle 8 (N=36) | Botulinum Toxin Type A 300U Treatment Cycle 9 (N=0) | Botulinum Toxin Type A 200U Treatment Cycle 9 (N=22) | Botulinum Toxin Type A 300U Treatment Cycle 10 (N=0) | Botulinum Toxin Type A 200U Treatment Cycle 10 (N=11) | Botulinum Toxin Type A 300U Treatment Cycle 11 (N=0) | Botulinum Toxin Type A 200U Treatment Cycle 11 (N=5) | Botulinum Toxin Type A 300U Treatment Cycle 12 (N=0) | Botulinum Toxin Type A 200U Treatment Cycle 12 (N=2) | Botulinum Toxin Type A 300U Treatment Cycle 13 (N=0) | Botulinum Toxin Type A 200U Treatment Cycle 13 (N=1)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrioventricular Block (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Umbilical Hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterocutaneous Fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adverse Drug Reaction (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 7 | 5 | 3 | 1 | 3 | 2 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium Difficile Colitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary Tract Infection Bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meningitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Necrotising Fasciitis (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Craniocerebral Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendon Rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Forearm Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Incisional Hernia (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine Cytology Abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foot Deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertebral Foraminal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/69 | 0/85 | 0/64 | 0/72 | 0/47 | 0/68 | 0/31 | 0/59 | 0/17 | 0/41 | 0/8 | 0/27 | 0/5 | 0/19 | 0 | 0/16 | 0 | 0/10 | 0 | 0/6 | 0 | 0/2 | 0 | 0 | 0 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thyroid Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Multiple Sclerosis Relapse (Nervous system disorders) | 4 | 4 | 4 | 0 | 3 | 3 | 4 | 2 | 1 | 1 | 0 | 3 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle Spasticity (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ischaemic Stroke (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myasthenia Gravis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mental Status Changes (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary Retention (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urethral Haemorrhage (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epididymitis (Reproductive system and breast disorders) | 0/69 | 1/85 | 0/64 | 0/72 | 0/47 | 1/68 | 1/31 | 0/59 | 0/17 | 0/41 | 0/8 | 0/27 | 0/5 | 0/19 | 0 | 0/16 | 0 | 0/10 | 0 | 0/6 | 0 | 0/2 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 2 | 4 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abortion Induced (Surgical and medical procedures) | 0/116 | 1/118 | 0/99 | 0/115 | 0/72 | 0/107 | 0/38 | 0/94 | 0/17 | 1/69 | 0/8 | 0/43 | 0/3 | 0/29 | 0 | 0/20 | 0 | 0/12 | 0 | 0/5 | 0 | 0/3 | 0 | 0/0 | 0 | 0/0
Angina Pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision Blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis Ischaemic (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large Intestine Perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Volvulus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device Dislocation (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema Peripheral (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis Acute (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Systemic Candida (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Localised Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tibia Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lupus-Like Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Multiple Sclerosis (Nervous system disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraparesis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute Psychosis (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stress Urinary Incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bladder Neck Obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urethral Stenosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic Prolapse (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral Ischaemia (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device Deployment Issue (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Impaired Healing (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaphylactic Reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abscess of Salivary Gland (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device Related Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint Dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous Cell Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional State (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neurogenic Bladder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erectile Dysfunction (Reproductive system and breast disorders) | 0/69 | 0/85 | 0/64 | 0/72 | 1/47 | 0/68 | 0/31 | 0/59 | 0/17 | 0/41 | 0/8 | 0/27 | 0/5 | 0/19 | 0 | 0/16 | 0 | 0/10 | 0 | 0/6 | 0 | 0/2 | 0 | 0 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral Vascular Disorder (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device Malfunction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Parotitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scar (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scrotal Haematoma (Injury, poisoning and procedural complications) | 0/69 | 0/85 | 0/64 | 0/72 | 0/4 | 0/68 | 1/31 | 0/59 | 0/17 | 0/41 | 0/8 | 0/27 | 0/5 | 0/19 | 0 | 0/16 | 0 | 0/10 | 0 | 0/6 | 0 | 0/2 | 0 | 0 | 0 | 0
Cervical Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cervical myelopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary Incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydroureter (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post Procedural Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Medical observation (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal Cord Compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mobility Decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/116 | 0/118 | 0/99 | 0/115 | 0/72 | 0/107 | 0/38 | 0/94 | 0/17 | 0/69 | 0/8 | 0/43 | 0/3 | 1/29 | 0 | 0/20 | 0 | 0/12 | 0 | 0/5 | 0 | 0/3 | 0 | 0/0 | 0 | 0/0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subcutaneous Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Botulinum Toxin Type A 300U Treatment Cycle 1 (N=185) | Botulinum Toxin Type A 200U Treatment Cycle 1 (N=203) | Botulinum Toxin Type A 300U Treatment Cycle 2 (N=163) | Botulinum Toxin Type A 200U Treatment Cycle 2 (N=187) | Botulinum Toxin Type A 300U Treatment Cycle 3 (N=119) | Botulinum Toxin Type A 200U Treatment Cycle 3 (N=175) | Botulinum Toxin Type A 300U Treatment Cycle 4 (N=69) | Botulinum Toxin Type A 200U Treatment Cycle 4 (N=153) | Botulinum Toxin Type A 300U Treatment Cycle 5 (N=34) | Botulinum Toxin Type A 200U Treatment Cycle 5 (N=110) | Botulinum Toxin Type A 300U Treatment Cycle 6 (N=16) | Botulinum Toxin Type A 200U Treatment Cycle 6 (N=70) | Botulinum Toxin Type A 300U Treatment Cycle 7 (N=8) | Botulinum Toxin Type A 200U Treatment Cycle 7 (N=48) | Botulinum Toxin Type A 300U Treatment Cycle 8 (N=0) | Botulinum Toxin Type A 200U Treatment Cycle 8 (N=36) | Botulinum Toxin Type A 300U Treatment Cycle 9 (N=0) | Botulinum Toxin Type A 200U Treatment Cycle 9 (N=22) | Botulinum Toxin Type A 300U Treatment Cycle 10 (N=0) | Botulinum Toxin Type A 200U Treatment Cycle 10 (N=11) | Botulinum Toxin Type A 300U Treatment Cycle 11 (N=0) | Botulinum Toxin Type A 200U Treatment Cycle 11 (N=5) | Botulinum Toxin Type A 300U Treatment Cycle 12 (N=0) | Botulinum Toxin Type A 200U Treatment Cycle 12 (N=2) | Botulinum Toxin Type A 300U Treatment Cycle 13 (N=0) | Botulinum Toxin Type A 200U Treatment Cycle 13 (N=0)
Diarrhoea (Gastrointestinal disorders) | 7 | 10 | 7 | 6 | 3 | 0 | 3 | 4 | 2 | 4 | 0 | 4 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema Peripheral (General disorders) | 6 | 8 | 3 | 3 | 4 | 6 | 3 | 2 | 2 | 1 | 0 | 2 | 0 | 2 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 100 | 118 | 86 | 92 | 61 | 84 | 28 | 60 | 11 | 35 | 4 | 21 | 3 | 15 | 0 | 12 | 0 | 7 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Muscle Spasticity (Nervous system disorders) | 4 | 1 | 2 | 3 | 1 | 0 | 1 | 1 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 5 | 6 | 3 | 5 | 3 | 0 | 1 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ovarian Cyst (Reproductive system and breast disorders) | 0/116 | 0/118 | 0/99 | 0/115 | 0/72 | 0/107 | 0/38 | 0/94 | 1/17 | 0/69 | 0/8 | 0/43 | 0/3 | 0/29 | 0 | 0/20 | 0 | 0/12 | 0 | 0/5 | 0 | 0/3 | 0 | 0/0 | 0 | 0
Urinary Retention (Renal and urinary disorders) | 42 | 41 | 13 | 15 | 8 | 11 | 0 | 4 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 10 | 9 | 7 | 5 | 6 | 1 | 1 | 3 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 6 | 13 | 4 | 6 | 3 | 4 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 4 | 17 | 5 | 4 | 2 | 4 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal Mycotic Infection (Infections and infestations) | 4/116 | 7/118 | 4/99 | 5/115 | 2/72 | 3/107 | 1/38 | 1/94 | 0/17 | 0/69 | 0/8 | 1/43 | 0/3 | 0/29 | 0 | 0/20 | 0 | 0/12 | 0 | 0/5 | 0 | 0/3 | 0 | 0/0 | 0 | 0
Expanded Disability Status Scale Score Increased (Investigations) | 7 | 10 | 13 | 12 | 4 | 8 | 2 | 5 | 0 | 3 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 5 | 8 | 10 | 8 | 2 | 6 | 2 | 0 | 0 | 2 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 5 | 6 | 7 | 6 | 1 | 9 | 2 | 5 | 0 | 4 | 0 | 3 | 0 | 3 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 7 | 6 | 3 | 2 | 0 | 10 | 1 | 2 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 5 | 2 | 1 | 4 | 1 | 2 | 1 | 3 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 3 | 1 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 8 | 7 | 2 | 3 | 1 | 1 | 1 | 0 | 3 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fracture Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hand Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes Zoster (Infections and infestations) | 1 | 1 | 0 | 1 | 3 | 1 | 1 | 2 | 0 | 2 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 5 | 10 | 3 | 5 | 5 | 4 | 1 | 7 | 0 | 4 | 0 | 1 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 2 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal Pruritus (Reproductive system and breast disorders) | 0/116 | 1/118 | 0/99 | 0/115 | 0/72 | 0/107 | 0/38 | 1/94 | 0/17 | 1/69 | 0/8 | 0/43 | 0/3 | 0/29 | 0 | 1/20 | 0 | 0/12 | 0 | 0/5 | 0 | 0/3 | 0 | 0/0 | 0 | 0
Bundle Branch Block Right (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Central Nervous System Function Test Abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fungal Skin Infection (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis Norovirus (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Osteomyelitis Acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Rhinitis Seasonal (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 4 | 5 | 2 | 0 | 0 | 2 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urine abnormality (Renal and urinary disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 8 | 9 | 3 | 4 | 3 | 4 | 1 | 1 | 1 | 3 | 0 | 2 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.